CLINICAL TRIAL: NCT05594875
Title: An Open-Label, Multi-Center Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of SHR-A1921 for Injection in Subjects With Advanced Solid Tumors
Brief Title: A Trial of SHR-A1921 for Injection in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1921-I-102-AUS
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: SHR-1921 single arm study in pt. with Advance solid tumors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1921 (Experimental)
  Interventions: Drug: SHR-1921

INTERVENTIONS:
Drug: SHR-1921 — Subject will receive a single dose of SHR-1921 at dose level 1/2/3 on Day of each cycles

SUMMARY:
The study is being conducted to evaluate the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of SHR-1921.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects consented and willing to provide required tumor tissue of sufficient quantity and of adequate tumor tissue content
3. Male or female
4. Subjects with clinically or pathologically confirmed advanced (recurrent, unresectable or metastatic) solid tumors who have failed prior standard of care therapy
5. ECOG performance status of 0-1

Exclusion Criteria:

1. Has uncontrolled clinically symptomatic pleural effusion, pericardial effusion, carcinomatous ascites
2. Has untreated brain metastasis, or with concomitant meningeal metastasis or spinal cord compression
3. Has known history of other documented malignancy
4. Has known history of acquired immunodeficiency syndrome (AIDS)
5. Has significant cardiovascular disease that is not well controlled, such as: (1) New York Heart Association (NYHA) Grade ≥ 2 cardiac failure
6. Has active or prior documented interstitial pneumonia/interstitial lung disease
7. Has experienced Grade ≥ 2 hemorrhage events within 4 weeks prior to the first dose
8. Has known active hepatitis B
9. Has known allergies to SHR-1921 component
10. Has other potential factors that may interfere with the study results, or result in the premature discontinuation as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | Screening up to study completion, an average of 1 year
  To check the numbers of AEs happened during the course of trial.
Number of subjects with laboratory tests findings of potential clinical importance | Screening up to study completion, an average of 1 year
  To check the Clinically significant and non clinically significant abnormal values during the course of trial.
Incidence of vital sign abnormalities e.g. Systolic and Diastolic BP, Pulse rate. | Screening up to study completion, an average of 1 year
  To measure the vital signs on regular basis for all study participants
Measure ECG | Screening up to study completion, an average of 1 year
  Number of subjects with clinically significant abnormal ECG QT Interval

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of SHR-1921 | Screening up to study completion, an average of 1 year
  To check what will be the maximum concentration participants will obtained of SHR-1921 in their blood plasma.
Area under the concentration-time curve (AUC 0-∞) from time 0 to infinity of SHR-1921 | Screening up to study completion, an average of 1 year
  To check the drug profile for absorption, distribution, metabolism and excretion for SHR-1921 in participants blood plasma
Time to Cmax (Tmax) of SHR-1921 | Screening up to study completion, an average of 1 year
  To check what time will it take to reach the maximum contraction of SHR-1921 in study participants
Clearance of SHR-1921 | Screening up to study completion, an average of 1 year
  The apparent clearance of SHR-1921(CL/F) of SHR-1921
Terminal elimination half-life (t1/2) of SHR-1921 | Screening up to study completion, an average of 1 year
  To check how much time SHR-1921 will take to eliminate half of it's concentration from participants.
Pharmacodynamics ("ADA" ) of SHR-1921. | Screening up to study completion, an average of 1 year
  To check the" Anti Drug Antibody" develops in participants against the SHR-1921 through blood sample

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Scientia Clinical Research, Sydney, New South Wales
  - Macquarie Hospital, Sydney, New South Wales
  - Sydney South West Private Hospital, Sydney, New South Wales
  - ICON Cancer Centre, Brisbane, Queensland